CLINICAL TRIAL: NCT00529087
Title: A Mulitcenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of Subcutaneous MOA-728 for the Treatment of Opioid-Induced Constipation in Subjects With Chronic Non-Malignant Pain
Brief Title: Study Evaluating Subcutaneous MOA-728 for the Treatment of Opioid-Induced Constipation (OIC) in Subjects With Chronic Non-Malignant Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3200K1-3356
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Results first posted 2010-05-11 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Constipation
Keywords: Opioid-Induced Constipation
MeSH Terms: conditions — Constipation; Opioid-Induced Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Other: placebo
- 2 (Experimental)
  Interventions: Drug: N-methylnaltrexone bromide (MOA-728)
- 3 (Experimental)
  Interventions: Drug: N-methylnaltrexone bromide (MOA-728)

INTERVENTIONS:
Drug: N-methylnaltrexone bromide (MOA-728) — Subcutaneous
  Arms: 2; 3
Other: placebo — placebo
  Arms: 1

SUMMARY:
The primary purpose of the protocol is to evaluate the safety, efficacy, and tolerability of subcutaneous MOA-728 versus placebo in subjects with chronic non-malignant pain who have Opioid-Induced Constipation (OIC).

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients with opioid-induced constipation and chronic non-malignant pain.
* Taking oral, transdermal, intravenous, or subcutaneous opioids.
* Willingness to discontinue all pre-study laxative therapy and use only study permitted rescue laxatives.

Exclusion Criteria

* History of chronic constipation before the initiation of opioid therapy.
* Other GI disorders known to affect bowel transit.
* Women who are pregnant, breast-feeding, or plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (72):
- United States (72):
  - Mobile, Alabama
  - Sun City, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Anaheim, California
  - Garden Grove, California
  - Hawaiian Gardens, California
  - Long Beach, California
  - Los Angeles, California
  - San Diego, California
  - Brandon, Florida
  - Cheifland, Florida
  - Clearwater, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Largo, Florida
  - Miami, Florida
  - Naples, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Spring Hill, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Stockbridge, Georgia
  - Chicago, Illinois
  - DeKalb, Illinois
  - Avon, Indiana
  - Indianapolis, Indiana
  - West Des Moines, Iowa
  - Shreveport, Louisiana
  - Sunset, Louisiana
  - Elkridge, Maryland
  - Boston, Massachusetts
  - Brockton, Massachusetts
  - Cadillac, Michigan
  - Paw Paw, Michigan
  - Traverse City, Michigan
  - Biloxi, Mississippi
  - Ocean Springs, Mississippi
  - Nixa, Missouri
  - Kalispell, Montana
  - Missoula, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Great Neck, New York
  - Valley Stream, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Dayton, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Levittown, Pennsylvania
  - Chattanooga, Tennessee
  - Austin, Texas
  - Beaumont, Texas
  - Colleyville, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Alexandria, Virginia
  - Christiansburg, Virginia
  - Hampton, Virginia
  - Spokane, Washington
  - Charleston, West Virginia

REFERENCES:
- [Derived] Liao SS, Slatkin NE, Stambler N. The Influence of Age on Central Effects of Methylnaltrexone in Patients with Opioid-Induced Constipation. Drugs Aging. 2021 Jun;38(6):503-511. doi: 10.1007/s40266-021-00850-w. Epub 2021 Mar 31. PMID 33788162
- [Derived] Michna E, Weil AJ, Duerden M, Schulman S, Wang W, Tzanis E, Zhang H, Yu D, Manley A, Randazzo B. Efficacy of subcutaneous methylnaltrexone in the treatment of opioid-induced constipation: a responder post hoc analysis. Pain Med. 2011 Aug;12(8):1223-30. doi: 10.1111/j.1526-4637.2011.01189.x. Epub 2011 Aug 2. PMID 21810165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide from August 2007 to September 2008.
Pre-assignment Details: Patients were screened up to 16 days.
Groups:
- MOA-728 QD (Double-blind): MOA-728 12 mg once daily (QD) for weeks 1 through 4
- MOA-728 QOD (Double-blind): MOA-728 12 mg once every other day, Placebo once daily on alternating days for weeks 1 through 4
- Placebo (Double-blind): Once daily for weeks 1 through 4
Period: Overall Study
Arm/Group | MOA-728 QD (Double-blind) | MOA-728 QOD (Double-blind) | Placebo (Double-blind)
Started | 150 | 148 | 162
Completed | 122 | 120 | 146
Not Completed | 28 | 28 | 16
Not completed — Adverse Event | 10 | 13 | 4
Not completed — Lost to Follow-up | 6 | 4 | 1
Not completed — Protocol Violation | 8 | 7 | 6
Not completed — Withdrawal by Subject | 3 | 3 | 3
Not completed — Protocol deviation | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MOA-728 QD (Double-blind) | MOA-728 QOD (Double-blind) | Placebo (Double-blind) | Total
Number analyzed (Participants) | 150 | 148 | 162 | 460
Age, Continuous [Mean (Standard Deviation); unit: years] — This baseline measure captures the double-blind population demographics in the arms MOA-728 QD, MOA-728 QOD and Placebo. It also captures the baseline demographics for the open-label portion of the study.
  years | 47.99 (10.74) | 48.64 (11.05) | 49.69 (10.77) | 48.79 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants] — This baseline measure captures the double-blind population demographics in the arms MOA-728 QD, MOA-728 QOD and Placebo. It also captures the baseline demographics for the open-label portion of the study
  Participants
    Female | 93 | 85 | 99 | 277
    Male | 57 | 63 | 63 | 183

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Having a Rescue-free Bowel Movement (RFBM) Within 4 Hours of the First Dose
Description: A rescue-free bowel movement was defined as a bowel movement where no laxatives were used during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone interactive voice response system (IVRS).
Time Frame: up to 4 hours
Population: Patients who were randomized and received at least 1 dose of double-blinded test article. For this analysis, the MOA-728 QD and MOA-728 QOD treatment groups were combined as the treatment regimen was the same through the first dose (day 1).
Measure: Number; unit: percentage of participants
Groups:
- MOA-728 QD and MOA-728 QOD: MOA-728 QD treatment group (12 mg every day) and MOA-728 QOD treatment group (12 mg once every other day, with placebo once daily on alternating days).
- Placebo: Once daily
Arm/Group | MOA-728 QD and MOA-728 QOD | Placebo
Number analyzed (Participants) | 298 | 162
percentage of participants | 34.2 | 9.9
Statistical Analysis 1: Comparison: MOA-728 QD and MOA-728 QOD vs Placebo; Test type: Superiority or Other; p < 0.001, Chi-squared; Treatment Difference = 24.4, 95% CI [17.3 to 31.4]

2. Primary Outcome: Percentage of Active Injections Resulting in Any Rescue-free Bowel Movement (RFBM) Within 4 Hours of Injection During the Double-blind Period
Description: A rescue-free bowel movement was defined as a bowel movement where no laxatives were used during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone interactive voice response system (IVRS). Active injections are those that contain study drug (e.g., daily injections in MOA-728 QD treatment group and every other injection for the MOA-728 QOD treatment group). The corresponding injections in the placebo group were used as controls.
Time Frame: 4 weeks
Population: Patients who were randomized and received at least 1 dose of double-blinded test article.
Measure: Mean (Standard Deviation); unit: percentage of active injections
Groups:
- MOA-728 QD: MOA-728 12 mg once daily (QD)
- MOA-728 QOD: MOA-728 12 mg once every other day (QOD), with placebo once daily on alternating days
- Placebo QD (Only QOD Injections): Placebo group using odd numbered injections corresponding to the active injections in the MOA-728 QOD group. The same placebo patients of 162 was used for each active drug group (QD and QOD).
- Placebo QD: Once daily
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo QD (Only QOD Injections) | Placebo QD
Number analyzed (Participants) | 150 | 148 | 162 | 162
percentage of active injections | 28.9 (26.2) | 30.2 (27.9) | 9.3 (12.6) | 9.4 (11.3)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Treatment Difference = 19.5, 95% CI [15.1 to 24.0]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo QD (Only QOD Injections); Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Treatment Difference = 20.9, 95% CI [16.1 to 25.7]

3. Secondary Outcome: Time to the First Rescue-free Bowel Movement (RFBM) After First Dose
Description: A rescue-free bowel movement was defined as a bowel movement where no laxatives were used during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone interactive voice response system (IVRS). Responses following first injection were censored at 24 hours or at time of the second injection, which ever occurred first.
Time Frame: up to 24 hours
Population: Patients who were randomized and received at least 1 dose of double-blinded test article.
Measure: Number; unit: % of subjects achieving RFBM in 24 hours
Groups:
- MOA-728 QD and MOA-728 QOD: MOA-728 12 mg once daily (QD) and MOA-728 12 mg once every other day (QOD), Placebo once daily on alternating days
Arm/Group | MOA-728 QD and MOA-728 QOD | Placebo
Number analyzed (Participants) | 298 | 162
% of subjects achieving RFBM in 24 hours | 46.0 (0.9) | 25.3 (0.5)
Statistical Analysis 1: Comparison: MOA-728 QD and MOA-728 QOD vs Placebo; Test type: Superiority or Other; p < 0.001, Log Rank; Log-rank test for comparisons of survival distributions

4. Secondary Outcome: Change From Baseline in Weekly Number of Rescue-free Bowel Movements (RFBM) for the Double-blind Period at 4 Weeks
Description: A rescue-free bowel movement defined as a bowel movement with no laxatives use during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were reported daily by patient using a telephone interactive voice response system (IVRS). The weekly number of RFBM was defined as the total number of RFBM reported during the double-blind period divided by the number of days the patient reported diary information in that period, and then multiplied by 7 to normalize to a weekly number.
Time Frame: Baseline and 4 weeks
Population: Patients who were randomized and received at least 1 dose of double-blinded test article. Last observation carried forward (LOCF).
Measure: Mean (Standard Error); unit: bowel movements
Groups:
- MOA-728 QOD: MOA-728 12 mg once every other day (QOD), Placebo once daily on alternating days
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
bowel movements | 3.1 (0.2) | 2.1 (0.2) | 1.5 (0.2)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Treatment as factor and baseline weekly RFBM as covariate; Treatment Difference = 1.6, 95% CI [1.1 to 2.1]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p = 0.011, ANCOVA; Treatment as factor and baseline weekly RFBM as covariate; Treatment Difference = 0.7, 95% CI [0.2 to 1.2]

5. Secondary Outcome: Weekly Number of Rescue-free Bowel Movements (RFBM) (Open-label Period)
Description: A rescue-free bowel movement was defined as a bowel movement where no laxatives were used during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone IVRS. The weekly number of RFBM was defined as the total number of RFBMs reported during study period divided by the number of days the patient reported diary information in that period, and then multiplied by 7 to normalize to a weekly number. Weekly number of RFBM determined as missing for <4 days of information.
Time Frame: 8 weeks
Population: Patients who continued into the open-label period and received at least 1 dose of test article. Observed case analysis.
Measure: Mean (Standard Deviation); unit: bowel movements
Groups:
- MOA-728 PRN (Open-label): MOA-728 12 mg as needed (PRN) during weeks 5 through 12
Arm/Group | MOA-728 PRN (Open-label)
Number analyzed (Participants) | 356
bowel movements | 3.7 (2.0)

6. Secondary Outcome: Percentage of Patients Achieving at Least 3 Rescue-free Bowel Movements (RFBM) Per Week in Double-blind Period
Description: A rescue-free bowel movement was defined as a bowel movement where no laxatives were used during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone IVRS. The weekly number of RFBM was defined as the total number of RFBM reported during the study week divided by the number of days the patient reported diary information in that period, and then multiplied by 7 to normalize to a weekly number.
Time Frame: 4 weeks
Population: Patients who were randomized and received at least 1 dose of double-blinded test article.
Measure: Number; unit: percentage of participants
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
percentage of participants | 58.7 | 45.3 | 38.3
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p < 0.001, Chi-squared; Treatment Difference = 20.4, 95% CI [9.5 to 31.3]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p = 0.212, Chi-squared; Treatment Difference = 7.0, 95% CI [-4.0 to 18.0]

7. Secondary Outcome: Percentage of Active Injections Resulting in Any Rescue-free Bowel Movement (RFBM) Within 1, 2, 3 and 6 Hour(s) in Double-blind Period
Description: as for outcome 2
Time Frame: Within 1-6 hours during 4 week double-blind period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of active injections
Groups:
- MOA-728 QOD: MOA-728 12 mg once every other day, Placebo once daily on alternating days
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo | Placebo QD (Only QOD Injections)
Number analyzed (Participants) | 150 | 148 | 162 | 162
percentage of active injections
  1 hour | 17.8 (21.1) | 17.3 (22.6) | 3.3 (5.5) | 3.2 (5.9)
  2 hours | 24.2 (24.7) | 24.1 (26.4) | 5.8 (8.5) | 5.4 (9.1)
  3 hours | 27.0 (25.8) | 28.0 (27.5) | 7.8 (9.9) | 7.5 (10.7)
  6 hours | 31.1 (26.1) | 32.5 (28.5) | 11.5 (13.1) | 11.1 (14.9)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; The statistical analysis for all time points (1, 2, 3 and 6 hours) is only shown once as the p value is the same for all time points; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo QD (Only QOD Injections); [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

8. Secondary Outcome: Percentage of Injections Resulting in Any Rescue-free Bowel Movement (RFBM) Within 1, 2, 3, 4 and 6 Hours in Double-blind Period
Description: as for outcome 1
Time Frame: Within 1-6 hours during 4-week double-blind period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of injections
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
percentage of injections
  1 hour | 17.8 (21.1) | 11.3 (15.3) | 3.3 (5.5)
  2 hours | 24.2 (24.7) | 16.2 (18.2) | 5.8 (8.5)
  3 hours | 27.0 (25.8) | 18.7 (18.8) | 7.8 (9.9)
  4 hours | 28.9 (26.2) | 20.4 (19.0) | 9.4 (11.3)
  6 hours | 31.1 (26.1) | 22.2 (19.3) | 11.5 (13.1)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; 1 hour; Test type: Superiority or Other; p < 0.001, ANOVA; Treatment as a factor; Mean Difference (Final Values) = 14.5, 95% CI [11.2 to 17.9]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; 1 hour; Test type: Superiority or Other; p < 0.001, ANOVA; Treatment as a factor; Mean Difference (Final Values) = 8.0, 95% CI [4.6 to 11.4]
Statistical Analysis 3: Comparison: MOA-728 QD vs Placebo; 2 hours; Test type: Superiority or Other; p < 0.001, ANOVA; Treatment as a factor; Mean Difference (Final Values) = 18.5, 95% CI [14.4 to 22.5]
Statistical Analysis 4: Comparison: MOA-728 QOD vs Placebo; 2 hours; Test type: Superiority or Other; p < 0.001, ANOVA; Treatment as a factor; Mean Difference (Final Values) = 10.4, 95% CI [6.3 to 14.5]
Statistical Analysis 5: Comparison: MOA-728 QD vs Placebo; 3 hours; Test type: Superiority or Other; p < 0.001, ANOVA; Treatment as a factor; Mean Difference (Final Values) = 19.3, 95% CI [15.0 to 23.5]
Statistical Analysis 6: Comparison: MOA-728 QOD vs Placebo; 3 hours; Test type: Superiority or Other; p < 0.001, ANOVA; Treatment as a factor; Mean Difference (Final Values) = 11.0, 95% CI [6.7 to 15.3]
Statistical Analysis 7: Comparison: MOA-728 QD vs Placebo; 4 hours; Test type: Superiority or Other; p < 0.001, ANOVA; Treatment as a factor; Mean Difference (Final Values) = 19.5, 95% CI [15.2 to 23.9]
Statistical Analysis 8: Comparison: MOA-728 QOD vs Placebo; 4 hours; Test type: Superiority or Other; p < 0.001, ANOVA; Treatment as a factor; Mean Difference (Final Values) = 11.0, 95% CI [6.6 to 15.4]
Statistical Analysis 9: Comparison: MOA-728 QD vs Placebo; 6 hours; Test type: Superiority or Other; p < 0.001, ANOVA; Treatment as a factor; Mean Difference (Final Values) = 19.7, 95% CI [15.2 to 24.1]
Statistical Analysis 10: Comparison: MOA-728 QOD vs Placebo; 6 hours; Test type: Superiority or Other; p < 0.001, ANOVA; Treatment as a factor; Mean Difference (Final Values) = 10.7, 95% CI [6.2 to 15.2]

9. Secondary Outcome: Percentage of Patients With a Weekly Rescue-free Bowel Movement (RFBM) Rate ≥ 3 and an Increase of at Least 1 in the Weekly RFBM Rate From Baseline for the Double-blind Period
Description: A rescue-free bowel movement was defined as a bowel movement where no laxatives were used during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone IVRS. The weekly RFBM rate was defined as the total number of RFBM reported during study period divided by the number of days the subject reported diary information in that period, and then multiplied by 7 to normalize to a weekly rate.
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
percentage of participants | 58.7 | 43.2 | 37.7
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p < 0.001, Chi-squared; Treatment Difference = 21.0, 95% CI [10.2 to 31.9]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p = 0.316, Chi-squared; Treatment Difference = 5.6, 95% CI [-5.3 to 16.5]

10. Secondary Outcome: Percentage of Patients With an Increase of at Least 1 in the Weekly Rescue-free Bowel Movement (RFBM) Rate From Baseline for the Double-blind Period at 4 Weeks
Description: as for outcome 9
Time Frame: Baseline and 4 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
percentage of participants | 74.7 | 68.2 | 54.9
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p < 0.001, Chi-squared; Treatment Difference = 19.7, 95% CI [9.4 to 30.1]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p = 0.016, Chi-squared; Treatment Difference = 13.3, 95% CI [2.6 to 24.0]

11. Secondary Outcome: Change in Weekly Number of Bowel Movements During Double-blind Period
Description: Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone interactive voice response system (IVRS). The weekly number of BM was defined as the total number of BMs reported during study period divided by the number of days the subject reported diary information in that period, and then multiplied by 7 to normalize to a weekly number.
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: bowel movements
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
bowel movements | 2.7 (0.2) | 1.7 (0.2) | 1.3 (0.2)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Treatment as factor, Baseline as covariate; Mean Difference (Final Values) = 1.4, 95% CI [1.0 to 1.9]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p = 0.102, ANCOVA; Treatment as factor, Baseline as covariate; Mean Difference (Final Values) = 0.4, 95% CI [-0.1 to 0.8]

12. Secondary Outcome: Change From Baseline in Weekly Number of Quality Rescue-free Bowel Movements (RFBM)
Description: RFBM defined as bowel movement with no laxatives during the prior 24 hours. Information on laxative use, bowel movements and assessments were reported daily by patient. Weekly number of quality RFBM was the total number of quality RFBM reported in study period divided by number of days with information and multiplied by 7 for a normalized weekly number. Stool quality assessed with the Bristol Stool Form Scale (7-points) (1=difficult to pass, 7=entirely liquid). A quality RFBM defined as one other than diarrhea (Bristol Type 1-5).
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: bowel movements
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
bowel movements | 2.4 (0.2) | 1.7 (0.2) | 1.3 (0.2)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Treatment Difference = 1.1, 95% CI [0.6 to 1.5]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Treatment Difference = 0.4, 95% CI [0.0 to 0.9]

13. Secondary Outcome: Change in Weekly Number of Complete Rescue-free Bowel Movements (RFBM)
Description: A rescue-free bowel movement defined as a bowel movement with no laxatives use during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were reported daily by patient using a telephone interactive voice response system (IVRS). Weekly number of complete RFBM was the total number of complete RFBM reported in study period divided by the number of days with information, and multiplied by 7 for a normalized weekly number. A complete RFBM has a sensation of complete evacuation.
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: bowel movements
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
bowel movements | 1.9 (0.1) | 1.2 (0.1) | 0.8 (0.1)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Treatment as factor, Baseline as covariate; Mean Difference (Final Values) = 1.2, 95% CI [0.8 to 1.6]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p = 0.012, ANCOVA; Treatment as factor, Baseline as covariate; Mean Difference (Final Values) = 0.5, 95% CI [0.1 to 0.9]

14. Secondary Outcome: Change in Bristol Stool Form Scale Score for Rescue-free Bowel Movements (RFBM)
Description: A rescue-free bowel movement was defined as a bowel movement where no laxatives were used during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone interactive voice response system (IVRS). The Bristol Stool Form Scale assessed stool quality using a 7-point scale, where Type 1 = separate hard lumps like nuts (difficult to pass) and Type 7 = watery, no solid pieces (entirely liquid.)
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
units on scale | 1.4 (0.1) | 1.2 (0.1) | 0.9 (0.1)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA; Treatment as factor, Baseline as covariate; Mean Difference (Final Values) = 0.5, 95% CI [0.2 to 0.7]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p = 0.119, ANCOVA; Treatment as factor, Baseline as covariate; Mean Difference (Final Values) = 0.2, 95% CI [-0.1 to 0.5]

15. Secondary Outcome: Change in Straining Scale Score of Rescue-free Bowel Movements (RFBM) From Baseline During Double-blind Period
Description: A rescue-free bowel movement was defined as a bowel movement where no laxatives were used during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone interactive voice response system (IVRS). The amount of straining associated with bowel movements was assessed using a 5-point straining scale, where 0=none and 4=very severe.
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
units on scale | -1.1 (0.1) | -1.1 (0.1) | -0.8 (0.1)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p = 0.008, ANCOVA; Treatment as factor, Baseline as covariate; Treatment Difference = -0.3, 95% CI [-0.5 to -0.1]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p = 0.015, ANCOVA; Treatment as factor, Baseline as covariate; Treatment Difference = -0.2, 95% CI [-0.5 to 0.0]

16. Secondary Outcome: Percentage of Patients With Improvement in Bristol Stool Form Scale Score for Rescue-free Bowel Movements (RFBM) by 1 Point During Open Label Period
Description: as for outcome 14
Time Frame: 8 weeks
Population: Patients who continued into the open-label period and received at least 1 dose of test article.
Measure: Number; unit: percentage of participants
Arm/Group | MOA-728 PRN (Open-label)
Number analyzed (Participants) | 361
percentage of participants | 57.9

17. Secondary Outcome: Percentage of Patients With Improvement in Straining Scale Score for Rescue-free Bowel Movements (RFBM) by 1 Point During Open Label Period
Description: as for outcome 15
Time Frame: 8 weeks
Population: Patients who continued into the open-label period and received at least 1 dose of test article.
Measure: Number; unit: percentage of participants
Arm/Group | MOA-728 PRN (Open-label)
Number analyzed (Participants) | 361
percentage of participants | 55.4

18. Secondary Outcome: Change in Percentage of Rescue-free Bowel Movements (RFBM) With Bristol Stool Form Scale in Type 3 or Type 4 From Baseline During Double-blind Period
Description: A rescue-free bowel movement was defined as a bowel movement where no laxatives were used during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone IVRS. The Bristol Stool Form Scale assessed stool quality using a 7-point scale, where Type 1=separate hard lumps like nuts (difficult to pass) and Type 7=watery, no solid pieces (entirely liquid.) Specifically, Type 3=like a sausage but with cracks on the surface, Type 4=Like a sausage or snake, smooth and soft.
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
percentage change | 18.7 (2.4) | 18.5 (2.4) | 17.6 (2.3)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p = 0.731, ANCOVA; Treatment as factor, Baseline as covariate; Mean Difference (Final Values) = 1.1, 95% CI [-5.4 to 7.7]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p = 0.779, ANCOVA; Treatment as factor, Baseline as covariate; Mean Difference (Final Values) = 0.9, 95% CI [-5.6 to 7.5]

19. Secondary Outcome: Change in Percentage of Rescue-free Bowel Movements (RFBM) Classified as Diarrhea or Watery Stools From Baseline During Double-blind Period
Description: A rescue-free bowel movement was defined as a bowel movement where no laxatives were used during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone interactive voice response system (IVRS). The Bristol Stool Form Scale assessed stool quality using a 7-point scale, where Type 1 = separate hard lumps like nuts (difficult to pass), Type 6 = fluffy pieces with ragged edges, a mushy stool, and Type 7 = watery, no solid pieces (entirely liquid.) This analysis included types 6 and 7.
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
percentage change | 11.7 (1.8) | 8.8 (1.8) | 6.1 (1.7)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p = 0.023, ANCOVA; Treatment as factor, baseline as covariate; Treatment Difference = 5.6, 95% CI [0.8 to 10.4]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p = 0.258, ANCOVA; Treatment as factor, baseline as covariate; Treatment Difference = 2.8, 95% CI [-2.0 to 7.6]

20. Secondary Outcome: Percentage of Patients With Any Diarrhea or Watery Rescue-free Bowel Movements (RFBM) During Open-label Period.
Description: as for outcome 19
Time Frame: weeks 5-12
Population: Patients who continued into the open-label period and received at least 1 dose of test article.
Measure: Number; unit: percentage of participants
Arm/Group | MOA-728 PRN (Open-label)
Number analyzed (Participants) | 361
percentage of participants | 50.1

21. Secondary Outcome: Change in Percentage of Rescue-free Bowel Movements (RFBM) With Straining Scale Scores of 0 or 1 (no, or Mild) From Baseline During Double-blind Period
Description: A rescue-free bowel movement was defined as a bowel movement where no laxatives were used during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone interactive voice response system (IVRS). The amount of straining associated with bowel movements was assessed using a 5-point straining scale, where 0=none, 1 = mild and 4=very severe.
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
percentage change | 31.5 (2.8) | 31.1 (2.8) | 24.5 (2.7)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p = 0.071, ANCOVA; Treatment as factor, baseline as covariate; Mean Difference (Final Values) = 7.0, 95% CI [-0.6 to 14.5]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p = 0.087, ANCOVA; Treatment as factor, baseline as covariate; Mean Difference (Final Values) = 6.6, 95% CI [-1.0 to 14.2]

22. Secondary Outcome: Change in Percentage of Rescue-free Bowel Movements (RFBM) With a Sensation of Complete Evacuation From Baseline During Double-blind Period
Description: A rescue-free bowel movement was defined as a bowel movement where no laxatives were used during the prior 24 hours. Information on laxative use, bowel movements and bowel movement assessments were self reported daily by the patient using a telephone interactive voice response system (IVRS). A complete RFBM has a sensation of complete evacuation.
Time Frame: 4 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | MOA-728 QD | MOA-728 QOD | Placebo
Number analyzed (Participants) | 150 | 148 | 162
percentage change | 27.4 (2.6) | 24.2 (2.6) | 19.9 (2.5)
Statistical Analysis 1: Comparison: MOA-728 QD vs Placebo; Test type: Superiority or Other; p = 0.038, ANCOVA; Treatment as factor, baseline as covariate; Mean Difference (Final Values) = 7.6, 95% CI [0.4 to 14.7]
Statistical Analysis 2: Comparison: MOA-728 QOD vs Placebo; Test type: Superiority or Other; p = 0.237, ANCOVA; Treatment as factor, baseline as covariate; Mean Difference (Final Values) = 4.3, 95% CI [-2.8 to 11.5]

ADVERSE EVENTS:
Groups:
- MOA-728 PRN (Open-label): MOA-728 12 mg as needed (PRN) for weeks 5 through 12
Arm/Group | MOA-728 QD (Double-blind) | MOA-728 QOD (Double-blind) | Placebo (Double-blind) | MOA-728 PRN (Open-label)
Serious Adverse Events (participants affected / at risk) | 5/150 | 1/148 | 2/162 | 4/364
Other Adverse Events (participants affected / at risk) | 74/150 | 67/148 | 62/162 | 137/364
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MOA-728 QD (Double-blind) (N=150) | MOA-728 QOD (Double-blind) (N=148) | Placebo (Double-blind) (N=162) | MOA-728 PRN (Open-label) (N=364)
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MOA-728 QD (Double-blind) (N=150) | MOA-728 QOD (Double-blind) (N=148) | Placebo (Double-blind) (N=162) | MOA-728 PRN (Open-label) (N=364)
Abdominal distension (Gastrointestinal disorders) | 1 | 3 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 29 | 23 | 6 | 26
Abdominal pain upper (Gastrointestinal disorders) | 2 | 8 | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 9 | 17 | 6 | 10
Flatulence (Gastrointestinal disorders) | 7 | 0 | 6 | 7
Nausea (Gastrointestinal disorders) | 13 | 17 | 10 | 15
Vomiting (Gastrointestinal disorders) | 1 | 11 | 8 | 5
Chills (General disorders) | 2 | 3 | 0 | 1
Feeling cold (General disorders) | 0 | 3 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 4 | 1 | 1
Oedema peripheral (General disorders) | 1 | 1 | 4 | 2
Urinary tract infection (Infections and infestations) | 2 | 3 | 2 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 7
Dizziness (Nervous system disorders) | 5 | 2 | 1 | 5
Headache (Nervous system disorders) | 6 | 5 | 4 | 9
Tremor (Nervous system disorders) | 2 | 5 | 1 | 3
Anxiety (Psychiatric disorders) | 3 | 3 | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 9 | 2 | 8
Piloerection (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 0
Hot flush (Vascular disorders) | 4 | 5 | 3 | 5
Orthostatic hypotension (Vascular disorders) | 3 | 1 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.